CLINICAL TRIAL: NCT03740581
Title: The Effect of Intensive Versus Conventional Glycemic Control in Diabetic Foot Ulcer Healing: a Randomised Control Trial
Brief Title: Intensive Versus Conventional Glycemic Control in Diabetic Foot Ulcer Healing
Acronym: InVeCoG:DFU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ashu Rastogi, Assistant Professor, Department of Endocrinology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGIMER ENDO
Record Dates: First submitted 2018-11-05; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic foot ulcer; Intensive glycemic control
MeSH Terms: conditions — Diabetic Foot | interventions — Insulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive (Active Comparator): New anti-diabetic drug regimen with (mandatory) Insulin >= 3 times per day
  Interventions: Drug: Insulin
- Conventional (No Intervention): Old anti-diabetic drug regimen with or without Insulin (<3 times per day) to be continued as before

INTERVENTIONS:
Drug: Insulin — Basal Bolus regimen (Participant to receive, Insulin >= 3 times per day)
  Arms: Intensive

SUMMARY:
Diabetic foot ulcer is one of the most serious, most costly and at times life threatening complication of diabetes. The lifetime incidence of foot ulcer occurrence in diabetes is up to 25%. Despite the advent of numerous types of wound dressings and off-loading mechanisms, the ulcer healing rates in diabetes have remained dismally low. Hyperglycemia impairs the inflammatory, proliferative and remodeling phases of an ulcer. There are retrospective studies linking improvement of HbA1c to wound area healing rate. The investigators hypothesised that intensive glycemic control in a patient of diabetic foot ulcer improves the healing process. To explore this hypothesis, the investigators are conducting this randomized control trial with the primary aim of wound healing in patients of diabetic foot ulcer on either intensive glycemic treatment or conventional (pre-existing) glycemic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Patients of DM according to ADA guidelines
3. HbA1c >8% and/or FBG >130 on 3 consecutive occasions
4. DFU: Wagner grade 2 & 3 or UTS 2-3B
5. Duration of ulcer <12 weeks
6. Wound size: >1cm2
7. Willingness to sign consent form & participate in the study
8. Capacity to attend visits at hospital for review

Exclusion Criteria:

1. Diagnosis with unpredictable healing ability e.g. malignancy, depression, HIV, CTD, steroid use
2. Dialysis requiring CKD & eGFR <30 ml/min
3. Active Charcot foot
4. PEDIS 4: life threatening DFU
5. Pregnancy
6. ABI <= 0.7
7. Refusal to give informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complete wound closure (epithelialisation) at 12 weeks in both intensive and conventional treatment groups. | 12 weeks
  Ulcer area to be measured by Wound Measurement Camera model WZ2.0 (bought from (Wound zoom incorporate, 2916, Borham Ave, Stevens Point, W1, USA 54481) at baseline, 4 and 12 weeks.

SECONDARY OUTCOMES:
Percent reduction in ulcer area (from baseline) at 4 & 12 weeks in both intensive and conventional treatment groups. | 4 and 12 weeks
  This will be calculated using the measured ulcer area for all participants, irrespective of wound closure status.
HbA1c at 4 & 12 weeks in both intensive and conventional groups. | 4 and 12 weeks
  This ill be done to correlate glycemic control with ulcer area at 4 and 12 weeks respectively.
Change in ulcer severity- Wagner and UTWSC classification. | 4 and 12 weeks
  Downgrade of ulcer severity based on two well established diabetic foot ulcer classification systems and there correlation with wound closure and glycemic control will be seen.
Incidence of any amputation. | 4 and 12 weeks
  This outcome to be correlated with the glycemic control in both the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Medical Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No